CLINICAL TRIAL: NCT03767010
Title: Implementation and Evaluation of a Perceptual Learning Module Aimed at Improving the Identification of the Brachial Plexus in the Interscalene Groove With Ultrasound
Brief Title: Implementation and Evaluation of a Perceptual Learning Module on the Identification of the Brachial Plexus
Acronym: MAP-IS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18.275
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Medical Education

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (no PLM) (Experimental): Control: Pre, post, delayed test Participants will not do the PLM, but will perform a pretest, a posttest and a delayed test at 6 months
  Interventions: Other: Control (no PLM)
- Experimental (PLM) (Experimental): Experimental: PLM group (pre, post, delayed test, PLM) Participants will do a pretest, the PLM, a posttest and a delayed test at 6 months
  Interventions: Other: PLM

INTERVENTIONS:
Other: Control (no PLM) — Pre, post, delayed test Participants will perform a pretest, a posttest and a delayed test at 6 months.
  Arms: Control (no PLM)
Other: PLM — PLM Participants will take the PLM on the location of the brachial plexus at the level of the interscalene groove on surface ultrasound images. They will also take a pretest, a post-test and a delayed test at 6 months. Pre, post, delayed test Participants will perform a pretest, a posttest and a delayed test at 6 months.
  Arms: Experimental (PLM)

SUMMARY:
Purpose:

This study is designed to:

1. Implement a website hosting perceptual learning modules (PLMs)
2. Implement and assess a PLM designed to improve the capacity of fourth-year medical students and first-year residents (novices) to locate the brachial plexus (BP) at the level of the interscalene groove on surface ultrasound images.

Hypothesis: The hypothesis of the study is that the PLM will improve the ability of novices to correctly locate the BP at the level of the interscalene groove on surface ultrasound images, compared to a control group.

DETAILED DESCRIPTION:
Introduction:

Regional anesthesia has greatly benefited in recent years from the use of ultrasound to facilitate the location of nerves and of their surrounding structures. Allowing real-time visualization of anatomical structures, ultrasound has been shown to improve the success rate of blocks, to decrease procedure times and to improve patient safety by reducing accidental injections into vessels and nerves.

Ultrasound-guided regional anesthesia training, however, remains a long process. The conventional way to develop expertise is to practice on patients. The learner does the techniques under the supervision of an expert, who gives him feedback. While well established, this approach has several limitations: In addition to being time-consuming, it is limited by the number of available cases and access to supervising experts.

Perceptual learning modules (PLMs) represent an alternative modality to teach image interpretation in regional anesthesia and are already used in other fields. PLMs are online tools created to enhance the development of pattern recognition, a skill required to efficiently interpret ultrasound-guided images. With PLMs, learners observe a series of images or videoclips and must answer a question about each image in a short period of time. Each answer is followed immediately by feedback (the correct answer). By observing a large number of images online and by receiving systematic and expert feedback, the trainee quickly learns to extract efficiently the required information from the image.

PLMs developed with real ultrasound images could complement current training methods in regional anesthesia. A PLM could be especially useful for learning the interscalene block. Identification of the BP in the interscalene groove is often difficult in the absence of a reliable vascular marker. Furthermore, the presence of important surrounding structures to be avoided, like the vertebral artery and the pleura, make accurate image interpretation crucial to avoid complications.

The aim of this study is to set up a PLM focusing on the location of the BP in the interscalene groove using ultrasound imaging. As a first step, ultrasound images of the neck of healthy volunteers will be collected. Subsequently, these images will be uploaded on a secured website and interpreted by experts. Finally, a study will be undertaken to test whether the PLM improves the ability of medical students and junior residents (novices) to correctly locate the brachial plexus in the interscalene groove using ultrasound images.

Methods:

Development of a website to host the new PLM from an already existing model

Two professional programmers collaborating with our team have already developed a website to host and evaluate another PLM. Using this site as a template, the same programmers will be responsible for creating a similar website for this project.

Acquisition of images in healthy volunteers

Each volunteer will correspond to a case and each case will consist of three elements:

1. A video of approximately thirty seconds of ultrasound images of the neck;
2. A video taken simultaneously showing the position of the operator's hand and of the ultrasound probe on the volunteer's neck as the ultrasound images shown in the first video are being acquired;
3. A static image corresponding to one of the last frames of the first clip.

Validation of cases by experts and construction of a case bank

1. Prior to inclusion in the study, the selected cases will be anonymized and uploaded to the website and then validated independently by 3 anesthesiologists who are experts in regional anesthesia;
2. For each case, each expert will have to circle the BP on the static image after viewing the simultaneous videos without time limitation;
3. For each case, in addition to identifying and locating the BP, the experts will have to rate the difficulty of identifying and locating the BP on a 4 point Likert scale.

Recruitment of volunteers will continue until a sufficient number of validated cases is available to build the PLM and two tests.

Development of the PLM (20 cases)

The PLM will be developed with validated cases distinct from those of the performance tests and will have the following characteristics:

1. For each case, both videos will play simultaneously and loop for up to 90 seconds;
2. A static image including the BP will also be displayed;
3. Participants will need to move a pointer over the static image and place it anywhere over what they think is the BP;
4. The website will then provide feedback to the participants: the BP will be highlighted on the static image for up to 30 seconds;
5. After the feedback, the following case will be presented.

Two blocks of 10 cases will be formed. These blocks will contain the same proportion of "easy" "moderate" and "hard" cases. Cases within a block will be shown in a random order, but participants will always see the two blocks in the same order.

Development and validation of two tests to assess the performance of learners (10 cases each)

The objective of the tests is different from that of the PLM since their purpose is to assess the ability of participants to correctly identify the BP at different points during the study. These tests will have the same format as the PLM, except that no expert feedback will be provided after each case.

Two test version will be created with different cases. The order of the cases within a test will be random.

Pilot study of the effect of PLM on learner performance

Fourth-year medical students and first-year residents in anesthesiology will be invited to participate via email. Consent will be given online. In the first session, participants will complete a short online questionnaire about their demographics and clinical experience with ultrasound-guided regional anesthesia. They will also be shown a short tutorial to familiarize them with the platform, with basic sonoanatomy of the neck, and with the ultrasound scanning technique.

Subsequently, they will be randomly assigned to one of two groups: Control Group or PLM Group. Both groups will participate in two on-line sessions. The project will proceed as follows according to the participant assignment group:

1. Control Group (tests only)

   * First 30-minute session, immediately after agreeing to participate in the study

     * pre-test (10 cases)
     * post-test (10 cases)
   * Second session lasting 15 minutes, 6 months after the first session

     * 6 months post-test (10 cases)
2. PLM Group (tests and PLM)

   * First session of 1h10, immediately after agreeing to participate in the study

     * pre-test (10 cases)
     * PLM (20 cases with feedback)
     * post-test (10 cases)
   * Second session lasting 15 minutes, 6 months after the first session

     * 6 months post-test (10 cases)

At the end of the study, participants of the Control group will be allowed to complete the PLM if they wish to.

ELIGIBILITY:
Inclusion Criteria:

* Fourth-year medical students and first-year residents having access to a computer with a high speed internet connection
* Fourth-year medical students and first-year residents with no significant experience in ultrasound-guided regional anesthesia

Exclusion Criteria:

* Smart phones and tablets will not be accepted due to their smaller screens.
* Significant experience with ultrasound-guided regional anesthesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Difference in correct locations of the BP between the pretest and the immediate post-test, for the Control group vs the PLM group. | At baseline (pretest) and on the immediate post-test
  The BP for a case will be considered correctly located if the participant has placed a pointer inside a predefined "target zone", determined as representing the BP by three independent regional anesthesia experts.

SECONDARY OUTCOMES:
Difference in the average distance of BP location | At baseline (pretest) and on the immediate post-test
  Difference in the average distance of the participant's pointer relative to the target zone between the pretest and the immediate post-test, for the Control group vs the PLM group.
Difference in correct locations of the BP | At baseline (pretest) and on the delayed test at 6 months
  Difference in correct locations of the BP between the pretest and the delayed post-test, for the Control group vs the PLM group.
Average response times during the various tests | At baseline (pretest), on an immediate post-test, and on the delayed test at 6 months
  This measure represents the fluency or automaticity with which images are interpreted, and can be used to evaluate the cognitive effort deployed to make a reading. Training not only allows the expert to make an accurate location. It also allows the expert to do it quickly, and therefore with little cognitive effort, an essential attribute in clinical practice.
For the PLM group only, the evolution of the participants' accuracy during the PLM | During the PLM, at the end of the first on-line session
  The change in the participants' rate of correct answers as they progress through the PLM; indeed, since learners will evaluate all case blocks in the same order, we can estimate an average learning curve for our population (pretest vs block 1 vs block 2 vs post-test)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Robitaille, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No